CLINICAL TRIAL: NCT07221578
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VQW-765 for the On-Demand Treatment of Acute Anxiety in Patients With Social Anxiety Disorder
Brief Title: Study to Evaluate the Efficacy and Safety of VQW-765 for the On-Demand Treatment of Social Anxiety Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VQW-765-3201
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: Social Anxiety Disorder; Social Phobia; SAD; Public Speaking Anxiety; Performance Anxiety
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VQW-765 (Experimental)
  Interventions: Drug: VQW-765
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VQW-765 — oral capsule
  Arms: VQW-765
Drug: Placebo — oral capsule
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of a single oral dose of VQW-765 compared to placebo in adults with social anxiety disorder.

DETAILED DESCRIPTION:
The study will enroll approximately 500 patients with current diagnosis of social anxiety disorder (SAD). Eligible participants will be randomly assigned to receive either a single oral dose of VQW-765 or placebo in a 1:1 ratio, followed by a psychosocial stress test. 1-2 weeks after the treatment visit, a safety follow-up assessment will be conducted remotely.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent.
2. Male and female subjects aged 18-65 years, inclusive.
3. Current diagnosis of social anxiety disorder.
4. Liebowitz Social Anxiety Scale total score ≥60.
5. Public Speaking Anxiety Scale total score ≥60.
6. Hamilton Depression Rating Scale score ≤18.

Exclusion Criteria:

1. Suicide attempts and/or suicidal ideation in the past 2 years or currently at risk of suicide in the opinion of the investigator.
2. History of bipolar disorder, schizophrenia, psychosis, seizures, delusional disorders, obsessive-compulsive disorder, or autism spectrum disorder.
3. Posttraumatic stress disorder or an eating disorder in the past 6 months.
4. Substance or alcohol use disorder in the past 6 months or positive in drug/alcohol screening.
5. Psychotherapy in the past 6 months.
6. Psychotropic medication in the past 2 months.
7. Current or planned pregnancy or nursing during the trial period.
8. Any other reason as determined by the Investigator which may lead to an unfavorable risk-benefit of study participation, or interference with study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | 1 day
  Subjective Units of Distress Scale (SUDS) during performance phase, scored from 0-100 with a higher score indicating higher distress.

SECONDARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | 1 day
  Subjective Units of Distress Scale (SUDS) during anticipation phase, scored from 0-100 with a higher score indicating higher distress.
State-Trait Anxiety Inventory - State Anxiety Scale (STAI-S) | 1 day
  State-Trait Anxiety Inventory - State Anxiety Scale (STAI-S), scored from 20 to 80 with higher scores indicating higher anxiety level.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 weeks
  Assessment of safety and tolerability of VQW-765, as measured by spontaneous reporting of adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Vanda Investigational Site, Phoenix, Arizona
  - Vanda Investigational Site, Scottsdale, Arizona
  - Vanda Investigational Site, Encino, California
  - Vanda Investigational Site, Newport Beach, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, San Jose, California
  - Vanda Investigational Site, Walnut Creek, California
  - Vanda Investigational Site, Denver, Colorado
  - Vanda Investigational Site, Jacksonville, Florida
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Orlando, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Suwanee, Georgia
  - Vanda Investigational Site, New Orleans, Louisiana
  - Vanda Investigational Site, Pikesville, Maryland
  - Vanda Investigational Site, Rockville, Maryland
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Princeton, New Jersey
  - Vanda Investigational Site, Albuquerque, New Mexico
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Charlotte, North Carolina
  - Vanda Investigational Site, Wilmington, North Carolina
  - Vanda Investigational Site, Moosic, Pennsylvania
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Orem, Utah

IPD SHARING:
Plan to Share IPD: No